CLINICAL TRIAL: NCT02451189
Title: RCT to Describe the Effects of Colon Delivered Acetate, Propionate and Butyrate on Satiety and Glucose Homeostasis
Acronym: PRO-ESTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scottish Universities Environmental Research Centre (Other)
Collaborators: NHS Greater Clyde and Glasgow (Other); University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Douglas Morrison, Senior Lecturer, Scottish Universities Environmental Research Centre
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO-ESTER STUDY
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Weight maintenance; Appetite; Energy intake; Dietary fibre; Short-chain fatty acids; Fermentation; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — inulin-propionate ester

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Inulin acetate ester (Experimental): Inulin acetate ester, 10g/day for 30 days
  Interventions: Dietary Supplement: Inulin acetate ester
- Inulin propionate ester (Experimental): Inulin propionate ester, 10g/day for 30 days
  Interventions: Dietary Supplement: Inulin propionate ester
- Inulin butyrate ester (Experimental): Inulin butyrate ester, 10g/day for 30 days
  Interventions: Dietary Supplement: Inulin butyrate ester

INTERVENTIONS:
Dietary Supplement: Inulin acetate ester — Inulin acetate ester supplementation (10g/d) for 30 days. Appetite measurements on day 15 and oral glucose tolerance test (OGTT) on day 30.
  Arms: Inulin acetate ester
Dietary Supplement: Inulin propionate ester — Inulin propionate ester supplementation (10g/d) for 30 days. Appetite measurements on day 15 and OGTT on day 30.
  Arms: Inulin propionate ester
Dietary Supplement: Inulin butyrate ester — Inulin butyrate ester supplementation (10g/d) for 30 days. Appetite measurements on day 15 and OGTT on day 30.
  Arms: Inulin butyrate ester

SUMMARY:
Obesity, with its associated co-morbidities, is a major public health challenge. It is estimated that by 2050, 60% of men and 50% of women will be clinically obese. Obesity is associated with increased risk of developing diabetes, cardiovascular disease, and certain cancers. The increasing epidemic of obesity has necessitated the study of the complex mechanisms underlying energy homeostasis. Food intake, energy balance and body weight are tightly regulated by the hypothalamus, brainstem and reward circuits, on the basis both of cognitive inputs and of diverse humoral and neuronal signals of nutritional status. Several gut hormones, including glucagon-like peptide-1 (GLP-1) and peptide YY3-36 (PYY), have been shown to play an important role in regulating short-term food intake. Peripheral administration of PYY or GLP-1 enhances satiety and reduces food intake in animals and man. PYY, GLP-1 along with a host of other hormones are produced by the gut in response to nutrient availability in different regions of the gut and provide an exquisite mechanism of nutrient sensing in response to dietary intake. These hormones therefore represent potential targets in the development of novel anti-obesity treatments. A novel and attractive strategy to induce appetite regulation is the enrichment of foods with components that stimulate the release of GLP-1 and PYY. The short chain fatty acids (SCFA) produced by microbial fermentation of dietary fibre in the colon have been shown to stimulate the release of PYY and GLP-1 from rodent enteroendocrine L cells, via stimulation of the G-protein coupled free fatty acid receptors (FFAR) on colonic L cells. However, it is not known whether the three SCFA, acetate, butyrate and propionate, differentially affect appetite and glucose control. The aim of this study is to compare the effects of increased colonic delivery of acetate, butyrate and propionate on appetite and glucose control in overweight men in a randomised crossover study.

DETAILED DESCRIPTION:
The role of SCFA in appetite regulation: SCFA have been shown to stimulate PYY and GLP-1 production in animal models and dietary fibre, of which SCFA are the major end products, induce appetite regulation in humans. However the evidence underpinning which dietary fibres induce appetite regulation in humans is very weak because of the difficulty in controlling studies with very high fibre intake. In a recent project funded under the BBSRC DRINC initiative (BB/H004815/1), the investigators have the first direct evidence that SCFA can directly regulate appetite in humans. Prior to this study, in order to achieve production of SCFA to a level, which is high enough to induce appetite-regulating effects, very large amounts of dietary fibre (>25 g/d and up to 40 g/d) are required, and compliance with high fibre diets is poor due to gastrointestinal side effects. Furthermore, supplementing diets with mixed high fibre does not predictably or reliably increase colonic SCFA production or circulating levels of SCFA in all human populations because of the variability in gut microbial activity. Finally, orally administered SCFAs are not palatable and are rapidly absorbed in the small intestine where L cells are sparse. In our studies to date we have focussed on the SCFA propionate because it has the highest affinity for the receptors and is an end product of metabolism in the microbiota and therefore seems the obvious target to manipulate to investigate the effects of SCFA on appetite regulation. To overcome the unpalatably high levels of fermentable dietary fibre needed to significantly increase colonic propionate levels, and the unpredictability in the production of the resulting SCFAs, the investigators have developed and tested a novel delivery system targeting the release of gram quantities of propionate in the proximal colon. It is estimated that the delivery system may lead to a 2-8 fold increase in colonic propionate, a level very difficult to achieve through feeding a mixed fermentable fibre diet. This level of propionate production might have been observed in ancestral diets and in parts of rural Africa where dietary fibre intake is very high. Previous work, conducted by the investigators, has also demonstrated that delivery system increases plasma propionate levels, reduces food intake in acute studies of appetite, and in a longer term study (24 weeks), positive effects on food intake, body composition, glucose homeostasis, circulating lipids, cholesterol and liver function, liver and visceral fat and weight management were observed. However, at present it is not known if acetate, propionate and butyrate exert similar effects on appetite and glucose metabolism. Therefore in this study we wish to compare the the effects of targeted delivery of acetate, propionate and butyrate to the proximal colon on appetite and glucose homeostasis in overweight men.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Healthy
* Overweight (BMI 25-40 kg/m2)

Exclusion Criteria:

* Weight change of > 3kg in the preceding 2 months
* Current smokers
* Substance abuse
* Excess alcohol intake
* Diabetes
* Cardiovascular disease
* Cancer
* Gastrointestinal disease
* Kidney disease
* Liver disease
* Pancreatitis
* Use of any medication except contraceptive pill
* Peri-menopausal
* Pregnancy
* Breastfeeding

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Energy intake at ad libitum meal | 8 hours
  Energy intake is measured at an ad libitum meal

SECONDARY OUTCOMES:
Subjective appetite sensations | 8 hours
  Appetite is rated on 100 mm visual analogue scales
Plasma glucose and insulin | 2 hours
  Oral glucose tolerance test: Fasting and 2h glucose and insulin concentrations following consumption of solution providing 75g glucose

OTHER OUTCOMES:
Intestinal bacteria composition | 24 hours
  Faecal samples will be collected to assess the impact of the NDC esters on gut bacteria composition
Lipids | 8 hours
  Serum triglycerides and cholesterol concentrations will be determined
Appetite regulating gut hormones | 8 hours
  Fasting and postprandial gut hormone concentrations will be measured
Liver function test | 1hour

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Morrison, PhD, Principal Investigator — Scottish Universitites Environmental Research Centre
Locations (1):
- Glasgow Clinical Research Facility, Glasgow, Lanarkshire, United Kingdom